CLINICAL TRIAL: NCT07283783
Title: INCLUDE Program: A Perioperative Wellness Program Tailored for Black Surgical Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202511072
Record Dates: First submitted 2025-12-04; First posted 2025-12-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Surgery
Keywords: Perioperative Care; Minority Mental Health; Anxiety; Depression; Polypharmacy; Behavioral Treatment; Medication Counseling; Coordination
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Health Promotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wellness Program for Perioperative Mental Health (Experimental): Enrolled participants will participate in the study for approximately 3 months after surgery. The participants will complete questionnaires at baseline, 1 month after surgery, and 3 months after surgery. The Wellness Program will consist of Cognitive Behavioral Therapy (CBT) and medication optimization.
  Interventions: Behavioral: Wellness Program

INTERVENTIONS:
Behavioral: Wellness Program — The BCBT intervention consists of 8 to 10 structured sessions delivered remotely via phone or Zoom, beginning in the preoperative period and continuing for approximately three months after surgery.
  The interventionist will offer a protocolized review of current medications with feedback as appropriate, under guidance by the study psychiatrist.
  As additional optional components of the Wellness Program, the study team will also offer faith-based counseling as well as the option to involve family and friends as active or passive participants in the program.

SUMMARY:
In this study, the investigators will evaluate the feasibility of the Wellness Program, including patient recruitment, screening and outcome measures, and feasibility of adapting the intervention with older Black surgical patients who endorse clinically significant symptoms of depression and/or anxiety.

ELIGIBILITY:
Inclusion Criteria Patients:

* Age ≥60 years
* Scheduled surgical procedure at BJH or BJWCH (oncologic, cardiac; orthopedic)
* Clinically significant depression or anxiety symptoms screened by the PHQ-ADS (Patient Health Questionnaire Anxiety and Depression Scale) ≥10
* Black or African American.

Exclusion Criteria Patients:

* Inability to provide informed consent;
* Severe cognitive impairment screened by the SBT (Short Blessed Test) ≥10
* Acutely suicidal
* Considered ineligible per the discretion of the surgeon or study PI
* Considered ineligible per the discretion of the surgeon or study PI

Caregiver participants:

If patients identify a caregiver that the patient would like to include in their Wellness Program, the caregiver will be invited to consent. Patients will provide contact information for their caregiver.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Reach of the study as measured by number of patients who agree to participate in the study out of total eligible to participate | Through completion of enrollment for all participants (estimated to be 9 months, time for participant 1 day)
Reach of the intervention as measured by number of patients who completed the intervention out of patients who agreed to participate in the study | Through completion of follow-up for all participants (estimated to be 12 months, time for participant 3 months)

SECONDARY OUTCOMES:
Percentage of instrument or data fields completed for Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) | Baseline, 1 month after surgery, and 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Abraham, Ph.D., FACMI, FAMIA, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after deidentification, will be available, upon request. In addition, the study protocol will be available upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers must provide a methodologically sound proposal that meets the approval of the author. Proposals should be directed to joannaa@wustl.edu. To gain access, data requestors will need to sign a data access agreement. Data will be available to the requestor indefinitely via encrypted e-mail service.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu